CLINICAL TRIAL: NCT02858102
Title: Impact From Aerobic Exercise (a Program of Physical Activity) in the Metabolic Syndrome, Neurocognition and Empowerment in Individuals With Severe Mental Disorders Including Depression, Bipolar Disorder and Psychosis: a Longitudinal Study
Brief Title: Impact of Aerobic Exercise on Metabolic Syndrome, Neurocognition and Empowerment in Individuals With Mental Disorders
Acronym: EXERTMG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundación Marques de Valdecilla (Other)
Collaborators: Centro de Investigación Biomédica en Red de Salud Mental (Network); Instituto de Investigación Marqués de Valdecilla (Other)
Responsible Party: Principal Investigator, Benedicto Crespo-Facorro, Associate Professor of Psychiatry, Fundación Marques de Valdecilla
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EXERTMG
Record Dates: First submitted 2016-08-03; First posted 2016-08-08 (Estimated); Last update posted 2020-02-07 (Actual); Status verified 2019-02

CONDITIONS: Metabolic Syndrome; Mental Disorders
Keywords: Schizophrenia; Psychosis; Obesity; Neurocognition; Depression; Bipolar disorder; Metabolomics; Biomarkers; Hypertension; Dyslipidemia; Hyperglycemia; Hypertriglyceridemia
MeSH Terms: conditions — Metabolic Syndrome; Mental Disorders; Schizophrenia; Psychotic Disorders; Obesity; Depression; Bipolar Disorder; Hypertension; Dyslipidemias; Hyperglycemia; Hypertriglyceridemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active treatment group (Active Comparator): Physical activity program: 36 sessions of physical activity lasting between 30-60 minutes for 12 weeks, three days per week.
  Interventions: Behavioral: Physical activity program
- Control group (No Intervention): No physical activity program

INTERVENTIONS:
Behavioral: Physical activity program — The intensity of physical activity will be adapted to the possibilities of the participants making individualized proposals to encourage participants to acquire active lifestyle habits to improve their health. All sessions end with a routine of relaxation and passive stretching. Simultaneously self-employment is controlled outside the guided sessions.
  Arms: Active treatment group

SUMMARY:
This study aims to develop a program of systematic physical exercise maintained for at least 12 weeks to normalize biomarkers of metabolic syndrome; improve neurocognition and social functioning; increase empowerment, self-esteem and self-efficacy and reduce self-stigma in individuals with severe mental disorder with metabolic syndrome.

DETAILED DESCRIPTION:
Major depressive disorder has an estimated annual prevalence of 4% in Spain and the risk of a major depressive episode is 10.6%. Although there are few studies available, there is growing evidence regarding the fact that patients with affective disorders have a higher morbidity and mortality in relation to general population. This mortality would be duplicated mainly due to suicides but also by other factors such as increased metabolic risk and cardiovascular diseases. In Europe, depression is one of the leading causes of lost productivity, early retirement and absence from work due to illness and it will be the first cause of disease burden worldwide in 2030 according to World Health Organization. Several reasons could explain it: from the adverse effects of medication, less access to health services, until unhealthy lifestyle options associated with a loss of quality of life related to health.

Bipolar disorder is a serious mental illness that can affect between 2 and 5% of the population. This disease has a major impact on patient functioning and it is in sixth place among all diseases as a global cause of disability. Depending on the studies, metabolic syndrome is present between 8 and 56% of patients with bipolar disorder what this leads to increased morbidity and mortality affecting of their quality of life.

Annual incidence rates of psychosis are from 0.2 to 0.4 per 1000 population and prevalence throughout life is about 1%, being similar between men and women although the start in women is later. The age of onset is between 15 and 30 years and it has a significant economic impact on patient, on his family and society in general. Schizophrenia is a psychotic disorder in which the person suffers from delusions or hallucinations with a disorganized thought or speech and negative symptoms that are not accompanied by insight. Historically it has been associated with greater vulnerability and higher rates of physical comorbidity and excess mortality. In physical comorbidity highlights cardiovascular diseases and they are attributed a 60% mortality together with metabolic syndrome, which is 2-3 times more frequent than in the general population. This increase in morbidity and mortality is related to a style of unhealthy life (bad eating habits and lack of exercise), use of antipsychotic drugs and disease as intrinsic factor.

There has been an increase in interest for the study of metabolic syndrome (MetS) in psychiatric patients in recent decades. Although his description has evolved over time, we can define the MetS as a group of risk factors (abdominal obesity, elevated blood pressure, elevated fasting plasma glucose, high serum triglycerides and low high-density lipoprotein (HDL cholesterol) levels) that predict the onset of coronary heart disease, type 2 diabetes, gallstones, asthma, sleep apnea, fatty liver disease and several cancers. The most commonly used criteria for his diagnosis are the National Cholesterol Education Program-Adult Treatment Panel III (NCEP-ATP III 2003), requires at least three of the following risk factors:

1. Elevated waist circumference: ≥102 cm in men and ≥88 cm in women.
2. Elevated serum triglycerides: ≥150 mg/dL or drug treatment.
3. Reduced HDL cholesterol: <40 mg/dL in men and <50 mg/dL in women or drug treatment.
4. Elevated blood pressure: systolic blood pressure ≥130 mm Hg or diastolic blood pressure ≥ 85 mm Hg or drug treatment.
5. Elevated fasting glucose: ≥100 mg/dL or drug treatment.

ELIGIBILITY:
Inclusion Criteria:

* Meeting Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) criteria for depression, bipolar disorder or psychosis (at least 5 years of diagnosis).
* Meet criteria for metabolic syndrome (NCEP-ATP III 2003).
* Capable of providing signed and dated written informed consent in accordance with Good Clinical Practice (GCP) and the local legislation.
* Women of child-bearing potential must be ready and able to use highly effective methods of birth control.

Exclusion Criteria:

* Dependence or severe alcohol consumers (>300 g/week).
* Co-infection with Hepatitis B, C or HIV.
* Cirrhosis diagnosed or presence of other hepatic comorbidities.
* Patients participating in a physical intervention program at least 6 months before inclusion.

Ages: 35 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-06 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Change in abdominal obesity measured by waist circumference | 6 months
  Abdominal obesity, also known as central obesity, is when excessive abdominal fat around the stomach and abdomen has built up to the extent that it is likely to have a negative impact on health.
  Men are considered to be at high risk from abdominal obesity if their waist measurements are 102 cm or higher, while women are considered to be at high risk if their waist measurements are 88 cm or higher.

SECONDARY OUTCOMES:
Change in dyslipidemia measured by serum triglycerides and/or high-density lipoprotein (HDL cholesterol) levels. | 6 months
  Dyslipidemia is an abnormal amount of lipids (e.g.,triglycerides, cholesterol and/or fat phospholipids) in the blood.
  The normal triglyceride level is between 30 and 150 mg/dL. The normal HDL cholesterol level is between 40 and 60 mg/dL.
Change in hypertension measured by blood pressure | 6 months
  Hypertension (HTN or HT), also known as high blood pressure (HBP), is a long term medical condition in which the blood pressure in the arteries is persistently elevated.
  Blood pressure is expressed by two measurements, the systolic and diastolic pressures, which are the maximum and minimum pressures, respectively. Normal blood pressure at rest is within the range of 100-130 millimeters mercury (mmHg) systolic and 60-85 mmHg diastolic.
Change in hyperglycemia measured by fasting plasma glucose | 6 months
  Hyperglycemia, or high blood sugar (also spelled hyperglycaemia) is a condition in which an excessive amount of glucose circulates in the blood plasma.
  A subject with a consistent range between 100-126 mg/dl is considered hyperglycemic, while above 126 mg/dl is generally held to have diabetes.
Effect of physical activity intervention on serum biomarkers by using metabolomics | 6 months
  Metabolomics can be defined as the quantitative and qualitative analysis of all metabolites (molecules with a molecular weight of less than 1,500 Da) in a given organism, resulting in the construction of a metabolome or metabolic fingerprint, analogous to the genome or the proteome. Metabolomics is based on high-resolution mass spectrometry coupled to ultra-performance liquid chromatography.
  The following biomarkers will be screened: Cytokines; Irisin, adiponutrin, adiponectin, resistin, leptin; Pro-inflammation status: tumor necrosis factor (TNF-a); Interleukin (IL-1b, IL-6), alpha-1-antitrypsin, serum amyloid A, fibrinogen, C reactive protein; Oxidative stress: LDL-oxidized and anti-LDL-oxidized antibodies.

CONTACTS AND LOCATIONS:
Overall Officials: Benedicto Crespo-Facorro, Professor, Principal Investigator — University Hospital Marqués de Valdecilla, IDIVAL, Department of Psychiatry, School of Medicine, University of Cantabria, Santander, Spain. CIBERSAM Centro Investigación Biomédica en Red Salud Mental, Madrid, Spain
Locations (1):
- University Hospital Marqués de Valdecilla, Santander, Cantabria, Spain

IPD SHARING:
Plan to Share IPD: No